CLINICAL TRIAL: NCT03018171
Title: Impact on Maternal and Fetal Wellbeing and on Labor Curve of Intrathecal Clonidine Addiction for Labor Analgesia. A Randomized Controlled Trial.
Brief Title: Intrathecal Clonidine Addiction for Combined Spinal Epidural Analgesia During Labor
Acronym: ICA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Giovanni Calibita Fatebenefratelli Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01.17
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Labor Pain
Keywords: clonidine, spinal injections
MeSH Terms: conditions — Labor Pain | interventions — Clonidine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- SC (Experimental): this arm will receive intrathecal clonidine addiction to sufentanil during combined spinal epidural analgesia for labor
  Interventions: Drug: Clonidine
- S (Active Comparator): this arm will receive intrathecal sufentanil during combined spinal epidural analgesia for labor
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Clonidine — Intrathecal clonidine addiction
  Arms: SC
Drug: Sufentanil — Intrathecal
  Arms: S

SUMMARY:
The study aims to evaluate the impact of the addition of 20 mcg of intrathecal clonidine in combined spinalepidural for labor analgesia on the local anesthetic consumption, on labor performance and on maternal fetal well-being.

ELIGIBILITY:
Inclusion Criteria:

* Written maternal informed consent
* Singleton pregnancy
* Gestational age ≥ 37 weeks,
* ASA I
* BMI < 30
* fetus in cephalic presentation

Exclusion Criteria:

* Suspect or certainty of fetal malformation,
* Presence of conditions such as preeclampsia, multiparity, preterm labor
* History of adverse reaction to α-2 adrenergic agonists
* Nicotine addiction
* Chronic use of opioid

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 268 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
local anesthetic consumption reduction | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Claroni, MD, Principal Investigator — Fatebenefratelli San Giovanni Calibita - Tiberine Island
Locations (1):
- San Giovanni Calibita Fatebenefratelli, Tiberine Island, Hospital, Rome, Italy